CLINICAL TRIAL: NCT05863897
Title: e-COGRAT: A Blended eHealth Intervention for Fatigue Following Acquired Brain Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Heliomare Revalidatie (Unknown)
Responsible Party: Principal Investigator, Aglaia Zedlitz, Assistant Professor, Universiteit Leiden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-COGRAT
Record Dates: First submitted 2023-04-14; First posted 2023-05-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Acquired Brain Injury; Fatigue
Keywords: Intervention; eHealth; Rehabilitation; Feasibility
MeSH Terms: conditions — Brain Injuries; Fatigue

STUDY DESIGN:
Intervention Model Description: A single-case experimental design with AB and follow-up phases across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eCOGRAT (Experimental)
  Interventions: Behavioral: e-COGRAT (a blended eHealth intervention)

INTERVENTIONS:
Behavioral: e-COGRAT (a blended eHealth intervention) — The blended eHealth intervention for fatigue complaints after ABI, e-COGRAT, is a cognitive behaviorial intervention. It consists of 12 weekly sessions, including 6 individual online sessions, 2 face-to-face group sessions and 4 online group sessions, in 4 groups of 4 patients.

SUMMARY:
Fatigue is a common, persistent consequence of acquired brain injury (ABI). Research into treatments that may alleviate post-ABI fatigue is been limited. Pharmacological treatment (methylphenidate) has shown the greatest scientific effects, but is complicated because the risk of adverse side effects and its potential for abuse. COGRAT, an evidence-based treatment combining cognitive therapy (CO) with graded activity training (GRAT), is found to be effective in treating fatigue in patients with acquired brain injury. However, therapist guided internet-based CBT (I-CBT) could offer a more accessible and cheaper alternative to this highly frequent face to face treatment. Moreover, I-CBT is found to be effective in a population with patients with psychiatric and chronic somatic disorders, including chronic fatigue syndrome. Recent studies suggests that I-CBT is effective for people with ABI as well. To obtain optimal benefit from both group delivered face to face therapy and e-health and to combine the available evidence of COGRAT and I-CBT in patients with ABI, we developed a blended e-health cognitive behavioral (group)intervention; e-COGRAT.

The goal of this intervention study is to evaluate the efficacy and feasibility of e-COGRAT to treat fatigue in people with ABI. The main questions it aims to answer are:

* Is a blended eHealth cognitive behavioral (group)intervention (e-COGRAT) effective as a treatment for fatigue in people with ABI?
* Is e-COGRAT the blended care variant of COGRAT, a cognitive behavioral group treatment for fatigue afer ABI, comparable to COGRAT in terms of efficacy?
* Will participants of e-COGRAT improve significant on overall fatigue, emotional well-being and participation?
* Will it be feasible for at least 80% of the participants to complete the intervention completely?

DETAILED DESCRIPTION:
A single case experimental design (SCED) with AB and follow-up phases across participants will be used. Within this study design, every participant will receive the blended eHealth cognitive behavioral (group)intervention (e-COGRAT). Patients who have given consent to participate in the study will be assigned to a treatment group by random assignment. Each group consists of 4 participants. Due to the group-based intervention all participants of each group will start simultaneously and immediately after baseline phase (2 weeks) with the 12-week intervention phase. Start dates will be predetermined based on the running dates of each group. The follow-up phase, immediately following after intervention phase, will take 24 weeks. The total duration of the study is 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* An ABI diagnosis (stroke and traumatic brain injury) in the chronic phase (≥6 months after injury)
* Complaints of severe fatigue (Checklist Individual Strength - subscale Fatigue score ≥ 40)
* Full comprehension of Dutch language
* Being cognitive capable of using the internet and having regular internet access.

Exclusion Criteria:

* Having severe cognitive deficits (Behavioural Assessment of the Dysexecutive Syndrome (BADS) < borderline)
* Having major untreated or unstable medical or psychiatric comorbidities (eg, epilepsy, psychosis)
* Patients with (complaints of) depression are excluded if the depression subscale of the Hospital Anxiety and Depression Scale (HADS) is > 10

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Daily fatigue | 1 year (daily in baseline and intervention phase and daily in the last week of follow-up)
  Primary outcome is the change in severity of fatigue complaints on a daily visual analogue scale (VAS) ("How would you rate your fatigue today?") which will be registered by text messages. Participants can indicate the severity of the experienced fatigue by given themselves a grade between 0 - 4. 0: "I'm not tired"; 1: "I'm a little bit tired"; 2: "tired"; 3: "pretty tired"; "; 4: "seriously tired". These grades will also be used in the intervention.

SECONDARY OUTCOMES:
Fatigue after ABI | 1 year (once in baseline, treatment and follow-up)
  Fatigue after ABI will be assessed with the Dutch Multifactor Fatigue Scale (DMFS). The DMFS measures 5 aspects of fatigue regarding the four weeks preceding the assessment: Impact of fatigue, Mental fatigue, Signs and Direct consequences of fatigue, Physical fatigue and Coping with fatigue. The DMFS contains 38 items. Questions are answered on a 5-point Likert scale. Subscales of the DMFS showed sufficient to good reliability (Cronbach's alpha = 0.70 to 0.91), good convergent validity with an existing fatigue scale, and good divergent validity with measures of mood and self-esteem.
Fatigue in the general population | 1 year (once in baseline, treatment and follow-up)
  Fatigue in the general population will be assessed with the Checklist Individual Strength - subscale Fatigue (CIS-f). The CIS-f contains 8 questions on fatigue severity regarding the two weeks preceding the assessment. The CIS-f has good reliability and is sensitive to change. Questions are answered on a 7-point Likert scale (1-7, higher scores represent higher fatigue).
Emotional distress | 1 year (once in baseline, treatment and follow-up)
  Depression and anxiety symptoms of the last week will be assessed with the Dutch version of the 14-item Hospital Anxiety and Depression Scale (HADS). The reliability of the HADS is good (Cronbach's Alpha = 0.71 to 0.90) as is the test-retest reliability (0.86-0.90) (Spinhoven et al., 1997). Questions are answered on a 4-point Likert scale (0-3): 7 items on the depression subscale (HADS-D) and 7 items of the anxiety subscale (HADS-A). Subscale sumscores are categorized as normal (0-7), mild (8-10), moderate (11-14) or severe (15-21).
Level of participation | 1 year (once in baseline, treatment and follow-up)
  The Utrecht Scale for Evaluation of Rehabilitation - Participation (USER-P) is a questionnaire to rate objective and subjective participation after rehabilitation. Internal consistency is satisfactory (Cronbach's Alpha = 0.70-0.91).
Feasibility of the overall online intervention | 1 year (once in treatment and follow-up)
  Feasibility will be assessed with structured interviews about overall usability, experienced benefits and difficulties and level of involvement. These interviews, for both participants and therapists, will take place posttreatment and after follow up.
Feasibility of each specific online session | 1 year (weekly during treatment and after follow-up)
  After each online session both patients and therapists fill in a questionnaire with questions about their experiences with the specific session concerning usability, content, lay out, potential technical difficulties and other assorted comments.

CONTACTS AND LOCATIONS:
Overall Officials: Aglaia M. Zedlitz, Dr., Study Chair — Leiden University
Locations (1):
- Heliomare, Wijk aan Zee, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zedlitz AM, Rietveld TC, Geurts AC, Fasotti L. Cognitive and graded activity training can alleviate persistent fatigue after stroke: a randomized, controlled trial. Stroke. 2012 Apr;43(4):1046-51. doi: 10.1161/STROKEAHA.111.632117. Epub 2012 Feb 2. PMID 22308241
- [Background] Visser-Keizer AC, Hogenkamp A, Westerhof-Evers HJ, Egberink IJ, Spikman JM. Dutch multifactor fatigue scale: a new scale to measure the different aspects of fatigue after acquired brain injury. Arch Phys Med Rehabil. 2015 Jun;96(6):1056-63. doi: 10.1016/j.apmr.2014.12.010. Epub 2015 Jan 2. PMID 25559057
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] van der Zee CH, Priesterbach AR, van der Dussen L, Kap A, Schepers VP, Visser-Meily JM, Post MW. Reproducibility of three self-report participation measures: The ICF Measure of Participation and Activities Screener, the Participation Scale, and the Utrecht Scale for Evaluation of Rehabilitation-Participation. J Rehabil Med. 2010 Sep;42(8):752-7. doi: 10.2340/16501977-0589. PMID 20809057
- [Background] Ali A, Morfin J, Mills J, Pasipanodya EC, Maas YJ, Huang E, Dirlikov B, Englander J, Zedlitz A. Fatigue After Traumatic Brain Injury: A Systematic Review. J Head Trauma Rehabil. 2022 Jul-Aug 01;37(4):E249-E257. doi: 10.1097/HTR.0000000000000710. Epub 2021 Aug 4. PMID 34354018
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Ford ME, Geurtsen GJ, Groet E, Rambaran Mishre RD, Van Bennekom CAM, Van Someren EJW. A blended eHealth intervention for insomnia following acquired brain injury: a randomised controlled trial. J Sleep Res. 2023 Feb;32(1):e13629. doi: 10.1111/jsr.13629. Epub 2022 May 31. PMID 35641443
- [Background] Theadom A, Barker-Collo S, Jones K, Dudley M, Vincent N, Feigin V. A pilot randomized controlled trial of on-line interventions to improve sleep quality in adults after mild or moderate traumatic brain injury. Clin Rehabil. 2018 May;32(5):619-629. doi: 10.1177/0269215517736671. Epub 2017 Oct 26. PMID 29072086
- [Background] van Beugen S, Ferwerda M, Hoeve D, Rovers MM, Spillekom-van Koulil S, van Middendorp H, Evers AW. Internet-based cognitive behavioral therapy for patients with chronic somatic conditions: a meta-analytic review. J Med Internet Res. 2014 Mar 27;16(3):e88. doi: 10.2196/jmir.2777. PMID 24675372
- [Background] Janse A, Worm-Smeitink M, Bleijenberg G, Donders R, Knoop H. Efficacy of web-based cognitive-behavioural therapy for chronic fatigue syndrome: randomised controlled trial. Br J Psychiatry. 2018 Feb;212(2):112-118. doi: 10.1192/bjp.2017.22. PMID 29436329